CLINICAL TRIAL: NCT01061619
Title: Pathway to Diagnosis of Ovarian Cancer: Observational Retrospective Multicenter Study
Brief Title: Pathway to Diagnosis of Ovarian Cancer
Acronym: MITO-12
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: MITO 12
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: prediagnostic symptoms; sentinel events; pathway to diagnosis
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the prediagnostic symptoms and the events along the pathway to diagnosis of women with ovarian cancer, referred for first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of ovarian cancer
* Indication for chemotherapy
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Previous chemotherapy
* Unable or unwilling to participate in interview

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of ovarian cancer, presenting for first-line chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-01; Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
the frequency and duration of symptoms in 12 months preceding ovarian cancer diagnosis | at baseline
time intervals in weeks between prediagnostic sentinel events (onset of persistent symptoms, first physician visit, diagnosis of ovarian cancer) | at baseline
description of prediagnostic patient experiences according to modified Andersen's model of 'total patient delay' | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Alessandro Morabito, M.D.,, Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli; Jane Bryce, MSN, Principal Investigator — National Cancer Institute, Naples; Marzia Falanga, BSN, Principal Investigator — S. Giuseppe Moscati Hospital, Avellino; Carmen Pisano, MD, Principal Investigator — National Cancer Institute, Naples; Marilina Piccirillo, MD, Principal Investigator — National Cancer Institute, Naples; Massimo Di Maio, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (30):
- UZ Leuven-Gynecological Oncology,, Leuven, Belgium
- Charité Universitätsmedizin Berlin Campus Virchow-Klinikum / Frauenklinik, Berlin, Germany
- Italy (28):
  - IRCCS Oncologico Bari, Oncologia Medica, Bari, BA
  - Ospedale Riuniti di Bergamo, U.O. di Ostetricia e Ginecologia, Bergamo, BG
  - Ospedale Fatebenefratelli, U.O. di Oncologia, Benevento, BN
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Università Cattolica del Sacro Cuore, Dipartimento di Oncologia, Campobasso, CB
  - Azienda Ospedaliera C. Poma, Mantova, MN
  - Azienda Ospedaliera V. Cervello, Palermo, PA
  - Ospedale S. Massimo, Day Hospital Oncologico, Penne, PE
  - Centro di Riferimento Oncologico, Divisione di Oncolgia Medica C, Aviano, PN
  - Ospedale S. Chiara, Trento, TN
  - Ospedale S. Bortolo ULSS 6, U.O. di Oncologia Medica, Vicenza, VI
  - Ospedale Mazzoni, Ascoli Piceno
  - Policlinico Universitario, Bari
  - Universita di Bari Policinico I Clinical Ostetrica e Ginecologica, Bari
  - Ospedale Fatebenefratelli, Benevento
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Universita Cattolica del Sacro Cuore, Campobasso
  - Ospedale A. Manzoni, Lecco
  - Istituto Nazionale Tumori, Milan
  - A.O. Univeristaria Policlinico, Modena
  - Azienda Ospedaliera D. Cotugno, Napoli
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli
  - Università Federico II, Cattedra di Oncologia Medica, Napoli
  - Ospedale Silvestrini, Perugia
  - Ospedale Civile S. Spirito, Pescara
  - A.O. S. Maria degli Angeli, Pordenone
  - Ospedale S. Giovanni Calibita Fatebenefratelli, UO di Oncologia, Roma
  - A.O. di Udine S. Maria della Misericordia, Udine